CLINICAL TRIAL: NCT06438575
Title: Point of Care Diagnosis of Vaginal Infections to Ensure Accurate Treatment: (PAT Study)
Brief Title: Point of Care Diagnosis of Vaginal Infections
Acronym: PAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharon L Hillier (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Sponsor-Investigator, Sharon L Hillier, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY24010118
Record Dates: First submitted 2024-05-24; First posted 2024-06-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Vaginitis; Bacterial Vaginosis; Yeast Vaginitis; Trichomonas Vaginitis
Keywords: Point-of-care diagnosis; Vaginitis; Symptomatic
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Trichomonas Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual Care (Other): Vaginitis diagnosis and treatment will be based on usual provider evaluation and treatment during the office visit
  Interventions: Diagnostic Test: Usual Care
- Same Day Results (Other): the Xpert® Xpress MVP test will be run in real time as a point of care test at the time of the office visit and the results will be made available to the provider in approximately one hour. Providers will be asked to use the MVP test result for diagnosis and treatment of the participant.
  Interventions: Diagnostic Test: Xpert® Xpress MVP test

INTERVENTIONS:
Diagnostic Test: Xpert® Xpress MVP test — The Xpert® Xpress MVP is an FDA-cleared point-of-care test for vaginitis diagnosis
  Arms: Same Day Results
Diagnostic Test: Usual Care — Usual methods used by the healthcare provider for vaginitis diagnosis
  Arms: Usual Care

SUMMARY:
Vaginal infections are a common gynecologic issue and may cause significant symptoms and discomfort for individuals. Point of care tests are used to diagnose infections in the office, with an advantage of quick diagnosis and treatment. Examples of point of care tests are urine pregnancy, rapid strep and COVID-19 tests. This study will enroll persons with vaginal complaints and compare diagnosis and treatment based on usual care to diagnosis and treatment using a Food and Drug Administration-approved point of care test for the diagnosis of vaginitis. The study is being done to better understand diagnosis, treatment, and satisfaction using point of care tests compared to usual care.

Participants will be randomized to one of two study arms:

Arm 1: the healthcare provider will perform their usual evaluation and tests to make the diagnosis and provide treatment, as needed.

Arm 2: the provider will be asked to use the results of the point-of-care test being used in the study to make the diagnosis and provide treatment, as needed.

Regardless of arm, all diagnoses and treatment will be provided through the healthcare provider. All participants will be contacted 2 weeks later to answer a questionnaire related to diagnosis, treatment, current symptoms, and satisfaction with their visit. Medical records related to vaginal complaints, up to 30 days from enrollment, will be reviewed by the study team to obtain information on symptoms, tests performed, results, and treatments prescribed.

DETAILED DESCRIPTION:
The goal of this randomized clinical trial is to evaluate whether same day testing using the Xpert® Xpress MVP test in a patient care setting results in a higher degree of appropriate treatment of vaginitis compared to standard of care for persons having vaginitis symptoms. Approximately 300 individuals who are complaining of vaginitis symptoms and are seeking care at one of the study participating offices within Magee-Womens Hospital will be invited to participate. In this study, the office visit will serve as the enrollment visit. After obtaining informed consent, participants will complete a brief questionnaire and self-collect three vaginal swabs for three tests that are FDA-cleared for vaginitis diagnosis: Xpert® Xpress MVP, BD MAX™ Vaginal Panel, and BD AffirmTM VPIII Microbial Identification Test. Participants will be randomized (1:1) into one of two arms after collecting swabs:

Arm 1, vaginitis diagnosis and treatment will be based on usual provider evaluation and treatment during the office visit. The Xpert® Xpress MVP test will be batched with delayed results made available to the provider following the participant's 2-week study follow-up telephone contact

. Arm 2, the Xpert® Xpress MVP test will be run in real time as a point of care test at the time of the office visit and the results will be made available to the provider in approximately one hour. Providers will be asked to use the MVP test result for diagnosis and treatment of the participant

All participants, regardless of arm, will complete a follow-up telephone contact approximately two weeks after their office visit to assess symptom resolution and satisfaction. Review and collection of electronic medical record information related to the office visit evaluation, testing, diagnosis and treatment will also be included.

A Healthcare Provider Sub study will also be performed. The sub study will include a baseline questionnaire completed by clinicians at participating offices and then a follow-up questionnaire administered to clinicians who provided care for at least one study participant. The sub study will help investigators understand how providers feel about point-of-care testing for vaginitis.

ELIGIBILITY:
Primary study

Inclusion Criteria:

* Complaining of at least one symptom of vaginitis: vaginal discharge, vaginal odor, vulvar or vaginal itch. Women having vulvar or vaginal discomfort such as irritation, burning, pain of less than 2 months duration are also eligible. Pregnant participants who complain of vaginal discharge will be required to have at least one additional vaginal symptom to be eligible.
* Seeking care at one of the participating offices.
* Able and willing to provide informed consent.
* Willing to undergo all study-related assessments and procedures, including self-collection of vaginal swabs, answering questions/surveys, agreeing to the review and collection of information from their medical record from the office (enrollment/index) visit and up to 4 weeks after the office visit.

Exclusion Criteria:

* Previous participation in this study.
* Any condition, that in the opinion of the investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Healthcare Provider Sub-study

Inclusion Criteria:

* Able and willing to provide informed consent
* Provided clinical care to at least one study participant on the date of their study enrollment
* Willing to undergo all study-related assessments including answering questions/surveys

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2024-06-16 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Number of participants prescribed appropriate treatment | Approximately 24 hours
  Number of participants prescribed appropriate treatment at index visit or within 24 hours of index visit. Appropriate treatment is defined as Centers For Disease Control recommended, or Food and Drug Administration approved treatment based on diagnosis from the self-collected samples.

SECONDARY OUTCOMES:
Number of participants that receive correct diagnosis of vaginitis | Approximately 2 weeks
  Number of participants whose vaginitis is correctly diagnosed by their healthcare provider. A positive result from both the Xpert® Xpress MVP and the BD MAX™ Vaginal Panel will be considered the gold standard for diagnosis of vaginitis/vaginosis.
Number of participants who experience resolution of vaginitis symptoms | Approximately 2 weeks
  Number of participants who experience resolution of vaginitis symptoms at the two week follow up contact assessed by participant's self-report.
Number of participants that are satisfied with their office visit | Approximately 2 weeks
  Number of participants that respond that they are satisfied or very satisfied with their diagnosis and treatment for vaginitis at the 2-week follow-up visit. Satisfaction is evaluated on a 5-point Likert scale with 1 being very satisfied and 5 being very dissatisfied.
Number of accurate BD AffirmTM VPIII test results | Approximately 2 weeks
  Number of participant samples for which the BD AffirmTM VPIII test results agree with the results from the gold standard, defined as a concordant positive or negative result from both the Xpert® Xpress MVP and the BD MAX™ Vaginal Panel.

OTHER OUTCOMES:
Number of healthcare providers that are satisfied with Xpert® Xpress MVP test | Approximately 14 months
  Number of healthcare providers that respond that they are satisfied or very satisfied with using the Xpert® Xpress MVP to diagnose and treat their patients' vaginitis. Satisfaction is evaluated on a 5-point Likert scale with 1 being very satisfied and 5 being very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillier SL, Austin M, Macio I, Meyn LA, Badway D, Beigi R. Diagnosis and Treatment of Vaginal Discharge Syndromes in Community Practice Settings. Clin Infect Dis. 2021 May 4;72(9):1538-1543. doi: 10.1093/cid/ciaa260. PMID 32350529
- [Background] Schwebke JR, Gaydos CA, Nyirjesy P, Paradis S, Kodsi S, Cooper CK. Diagnostic Performance of a Molecular Test versus Clinician Assessment of Vaginitis. J Clin Microbiol. 2018 May 25;56(6):e00252-18. doi: 10.1128/JCM.00252-18. Print 2018 Jun. PMID 29643195
- [Background] Wiesenfeld HC, Macio I. The infrequent use of office-based diagnostic tests for vaginitis. Am J Obstet Gynecol. 1999 Jul;181(1):39-41. doi: 10.1016/s0002-9378(99)70433-3. PMID 10411793